CLINICAL TRIAL: NCT01852253
Title: Clinical and Microbiological Evaluation Implant Surface Decontamination With 2% Chlorhexidine in the Surgical Treatment of Peri-implantitis; a Double Blind Controlled Randomized Clinical Study
Brief Title: Implant Surface Decontamination With 2 % Chlorhexidine in Peri-implantitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31262.042.10
Record Dates: First submitted 2013-05-03; First posted 2013-05-13 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases; Peri-implantitis
Keywords: Dental implants; Periodontal diseases; Peri-implantitis; Chlorhexidine; Microbiology
MeSH Terms: conditions — Periodontal Diseases; Peri-Implantitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% chlorhexidine (Active Comparator): Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline and 1 minute of local application of a 2 % chlorhexidine solution. After 1 minute of saline rinsing the gingival flap will be returned slightly apical (in order to reduce pockets) and will be firmly sutured. The surgery is followed by 2 weeks of rinsing with 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol twice daily during 30 seconds.
  Interventions: Procedure: 2% chlorhexidine
- 0.12% chlorhexidine (Sham Comparator): Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline and 1 minute of local application of a 0.12 % chlorhexidine solution. After 1 minute of saline rinsing the gingival flap will be returned slightly apical (in order to reduce pockets) and will be firmly sutured. The surgery is followed by 2 weeks of rinsing with 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol twice daily during 30 seconds.
  Interventions: Procedure: 0.12% chlorhexidine

INTERVENTIONS:
Procedure: 2% chlorhexidine
  Arms: 2% chlorhexidine
Procedure: 0.12% chlorhexidine
  Arms: 0.12% chlorhexidine

SUMMARY:
Peri-implantitis is a infectious disease that resides in the mucosa surrounding dental implants and also affects the supporting bone. Because the number of implants placed in everyday clinical practice is continuously increasing, is it reasonable to anticipate an increasing prevalence of peri-implantitis. This underlines the necessity for a predictable therapy. However, from the literature there is very little reliable evidence suggesting which could be the most effective interventions for treating periimplantitis.

The primary objective of this controlled clinical study is to evaluate the clinical effect of decontamination of the implant surface during the surgical treatment of peri-implantitis using a 2% chlorhexidine solution or a 0.12% chlorhexidine solution. The secondary objective is to assess the microbiological effect of decontamination of the implant surface during the surgical treatment of peri-implantitis using a 2% chlorhexidine solution or a 0.12% chlorhexidine solution.

The primary study parameter is the change from baseline in modified bleeding index. Secondary study parameters are: change in microbial composition of the biofilm covering the dental implant surface; microbiological composition of the peri-implant sulcus; change in probing pocket depth;change in suppuration on probing; change in radiographic marginal bone level on standardized intraoral radiographs; change in modified plaque index; implant failure, defined as implant mobility of previously clinically osseointegrated implants and removal of non-mobile implants because of progressive marginal bone loss or infection; complications and adverse events. It is hypothesized that decontamination of the implant surface with 2% chlorhexidine leads to a greater decrease in modified bleeding index than decontamination with a 0.12% chlorhexidine solution.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age;
* The patient has at least one endosseous implant in the oral cavity with clinical and radiographical signs of peri-implantitis. Peri-implantitis is defined as a loss of marginal bone more than or equal to 2 mm as compared to a fixed reference point on the dental implant, in combination with bleeding and/or suppuration on probing and a peri-implant probing depth more than or equal to 5 mm;
* The implants have been exposed to the oral environment for at least two years;
* The patient is capable of understanding and giving informed consent.

Exclusion Criteria:

* Medical and general contraindications for the surgical procedures;
* A history of local radiotherapy to the head and neck region;
* Pregnancy and lactation;
* Insulin dependent diabetes;
* Systemic use of antibiotics during the last 2 months;
* Long-term use of anti-inflammatory drugs;
* Incapability of performing basal oral hygiene measures as a result of physical or mental disorders;
* Active, uncontrolled periodontal pathology of the remaining dentition;
* Local use of antibiotics or use of other anti-septic / antimicrobial therapies in the oral cavity during the last 2 months;
* Bruxism;
* Implants placed in skin grafted areas;
* Implants with bone loss due to other reasons than bacterial infection (e.g. loose screw, inadequate positioning of the implant);
* Implants with bone loss exceeding 2/3 of the length of the implant or implants with bone loss beyond the transverse openings in hollow implants;
* Implant mobility;
* Implants at which no position can be identified where proper probing measurements can be performed;
* Previous surgical treatment of the peri-implantitis lesions;
* Previous non-surgical treatment of the peri-implantitis lesions during the last 6 months (scaling or curettage).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in modified bleeding index. | baseline, 3, 6 and 12 months after treatment

SECONDARY OUTCOMES:
Change in microbial composition of the biofilm covering the dental implant surface | during treatment: 'after granulation tissue removal' and 'after mechanical and chemical decontamination procedure'
Microbiological composition of the peri-implant sulcus | before treatment and 3, 6 and 12 months after treatment
Change from baseline in probing pocket depth | baseline and 3, 6 and 12 months after treatment
Change from baseline in suppuration on probing | baseline and 3, 6 and 12 months after treatment
Change from baseline in radiographic marginal bone level on standardized intraoral radiographs | baseline and 3, 6 and 12 months after treatment
Change from baseline in modified plaque index | baseline and 3, 6 and 12 months after treatment
Implant failure, defined as implant mobility of previously clinically osseointegrated implants and removal of non-mobile implants because of progressive marginal bone loss or infection | 3, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] de Waal YC, Raghoebar GM, Huddleston Slater JJ, Meijer HJ, Winkel EG, van Winkelhoff AJ. Implant decontamination during surgical peri-implantitis treatment: a randomized, double-blind, placebo-controlled trial. J Clin Periodontol. 2013 Feb;40(2):186-95. doi: 10.1111/jcpe.12034. Epub 2012 Dec 4. PMID 23211012
- [Derived] de Waal YC, Raghoebar GM, Meijer HJ, Winkel EG, van Winkelhoff AJ. Implant decontamination with 2% chlorhexidine during surgical peri-implantitis treatment: a randomized, double-blind, controlled trial. Clin Oral Implants Res. 2015 Sep;26(9):1015-23. doi: 10.1111/clr.12419. Epub 2014 May 26. PMID 24861411